CLINICAL TRIAL: NCT02925754
Title: Catastrophism Among Chronic Pain Patients in Rheumatology
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2015/CGV-04
Record Dates: First submitted 2016-09-16; First posted 2016-10-06 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-09

CONDITIONS: Catastrophizing Pain

STUDY DESIGN:
Time Perspective: Cross-Sectional

SUMMARY:
Pain catastrophizing is conceptualized as a negative cognitive-affective response to anticipated or actual pain and has been associated with a number of important pain-related outcomes.

The aims of this study are

1. To describe the characteristics of the patients and determinants of catastrophizing in chronic painful patients hospitalized in rheumatology in the Nîmes University Hospital
2. To describe the impact of the catastrophizing on the level of insomnia and the drugs consumption in chronic painful patients hospitalized in rheumatology in the Nîmes University Hospital

ELIGIBILITY:
Inclusion Criteria:

* adults hospitalized in the department of rheumatology of the Nîmes University Hospital with chronic pain (≥ 6 months)

Exclusion Criteria:

* benzodiazepine or neuroleptic use for epilepsia, alcool, psychiatric disorders
* Restless Legs syndrom
* Obstructive Sleep Apnea
* narcolepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults hospitalized in the department of rheumatology of the Nîmes University Hospital with chronic pain (≥ 6 months)
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2015-08; Primary Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Pain Catastrophizing Scale | Day 0